CLINICAL TRIAL: NCT04097990
Title: Characterization of Fatty Acid Composition of Triglycerides in Patients With Hypertriglyceridemia-induced Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Rom Keshet, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6390-19-SMC
Record Dates: First submitted 2019-09-09; First posted 2019-09-20 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 10 healthy participants, 10 participants with hypertriglyceridemia without prior pancreatitis and 10 participants with hypertriglyceridemia and at least one case of severe pancreatitis in the last 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy participants (Other): healthy participants
  Interventions: Other: blood sample
- hypertriglyceridemia without prior pancreatit (Other)
  Interventions: Other: blood sample
- hypertriglyceridemia and at least one case of (Other)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — a 5 cc blood sample will be taken after a 12-hour fast for separation of triglycerides from the serum and for checking fatty acid levels

SUMMARY:
) Finding a unique pattern in the triglyceride composition of patients with hypertriglyceridemia that increases the chances of getting pancreatitis and which can serve as a laboratory predictive tool for patients and define them as a at-risk population.

2) Finding the typical fatty acid composition in triglycerides for patients at high risk of pancreatic acute inflammation that can be used to develop unique drugs for pancreatic acute inflammation caused by high levels of triglycerides.

DETAILED DESCRIPTION:
The study will be conducted at the Sheba Medical Center Lipid Institute, number of participants: 10 healthy participants, 10 participants with hypertriglyceridemia without prior pancreatitis and 10 participants with hypertriglyceridemia and at least one case of severe pancreatitis in the last 5 years.

A total of 30 participants Participants who are found suitable during their visit to the Lipid Institute Clinic or during their hospitalization at Sheba Medical Center will receive an explanation of the study, will be asked to sign a consent form. And check the fatty acid levels. Healthy volunteers who meet the inclusion conditions will also be asked to sign a consent form and their blood will be taken and kept frozen for further study

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy participants - triglyceride levels< 150 mg / dl over the past 5 years, with no diabetes or cardiovascular disease in the background.

  2) Participants with triglyceride levels 1000-5000 mg / dl without acute pancreatitis cases in the past.

  3) Participants with triglyceride levels 1000-5000 mg / dL and at least one case of acute pancreatitis in the last 5 years.

Exclusion Criteria:

1. A past pancreatitis event that occurred with measurement of triglyceride levels greater than 5000 mg / dL.
2. Acute pancreatitis events in the past that occurred for a cause other than hypertriglyceridemia -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Finding a unique pattern in the triglyceride composition | one year
  Fatty acids will be analyzed in a gas-chromatographer and their concentration in plasma will be measured by comparison to a known-consentration standard fatty acid solution. Concentration will be presented as mg/dL (miligrams per deciliter) or as a fold change concentration relative to the concentration in plasma of control subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Lipid center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No
Absolute medical confidentiality will be kept on all participants' details. All details will be kept locked while the tests containing the participants' blood or the biological materials produced from it will be marked in serial numbers only.